CLINICAL TRIAL: NCT06826638
Title: Investigate Neuro-rehabilitation Active Ingredients of Specific Task-oriented Training In People With Multiple Sclerosis With Different Challenging Conditions and Extrinsic Feedbacks
Brief Title: Unraveling Active Ingredients of Neurorehabilitation: Investigating Cortical Activity During Task-oriented Exercises
Acronym: INSIDE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Università degli Studi of Genova (Unknown); University of Milan (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/R-Multi/021
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Healthy Volunteer
Keywords: rehabilitation; multiple sclerosis; motor control; cortical plasticity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple sclerosis: A sample of 20 consecutive PwMS will be recruited.
- Healthy volunteers: We will recruit a group of healthy individuals to obtain normative reference data. These individuals will be matched for sex and age with the subjects having multiple sclerosis.

SUMMARY:
The driving idea of this project is to use new imaging techniques during 0functional movements to study relearning during a typical rehabilitation session.

The novelty of this project is to move from studies inquiring changes in brain activity patterns before and after rehabilitation toward a paradigm in which cortical activity is studied during the execution of the exercise. This would allow better understanding of cortical mechanisms underpinning functional improvements.

The project builds on preceding studies, partially funded by FISM, from the three research units involved in this project, aimed at assessing the impact of rehabilitation on mobility and balance and at assessing the effects of neurorehabilitation on brain plasticity. In this study, we will include 40 healthy subjects and a sample of 20 consecutive People with Multiple Sclerosis (PwMS), and we will investigate brain cortical activity during a typical session of task-oriented exercises. In specific, participants will undergo a treadmill training in which they will be required to keep their trunk and head stable in space using a biofeedback device. To study the effects of the session in improving dynamic stability, Head/trunk movements will be registered by inertial measurement units, while cortical activity will be concurrently assessed by functional near-infrared spectroscopy (fNIRS).

The first phase of the project will include healthy subjects and will be useful to understand the main cortical areas involved in the proposed motor tasks, in order to design the appropriate montage and protocol for fNIRS acquisition in PwMS. Finally, the analysis of the possible differences in cortical activation during different experimental conditions (e.g., biofeedback rehabilitation) in healthy subjects and PwMS will serve to develop a model for neurological rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* subjects between 18 and 60 years of age,
* diagnosis of MS (McDonald criteria, Thompson et al, 2018), stable disease course without worsening more than 1 EDSS point over the last 3 months, EDSS between 3 and 4.5 points,
* healthy right-handed volunteers,
* able to release a written informed consent.

Exclusion Criteria:

* Unable to comprehend the aims of the study and to follow test instructions;
* Diagnosis of major depression (DSM-5);
* Severe joint and/or bone disorders interfering with balance and gait (based upon clinical judgment);
* Cardiovascular diseases;
* Severe visual impairments interfering with the execution of the protocol;
* epilepsy;
* intake of neuroleptic and antiepileptic drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People with Multiple sclerosis people affiliated with the rehabilitation center of the IRCCS Santa Maria Nascente of the Don Gnocchi Foundation will be recruited. Participants should be able to maintain upright posture without any assistance for 30 seconds, and to walk without any assistance.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Head and trunk movements quantified with Inertial Measurement Units (IMU) | Baseline
  The following variables are calculated: (1) the angular displacements in the sagittal and frontal planes, calculated as 1 standard deviation (SD) from the angular displacement data; and the head and angular velocities, which are the root mean square of the first derivative of angular displacements in the sagittal and frontal planes.
Cortical activation with Functional Infrared Spettroscopy (fNIRS) | Baseline
  fNIRS data analysis will identify the acquisition channels (and hence the cortical areas) significantly active in the different experimental conditions.

SECONDARY OUTCOMES:
10 Meters walking test | Baseline
  The 10-Meter Walking Test (10MWT) is a commonly used assessment to measure walking speed and functional mobility, especially in individuals with neurological conditions like multiple sclerosis
Twelve-Item Multiple Sclerosis Walking Scale (MSWS_12) | Baseline
  to assess walking perceived ability of people with multiple sclerosis. The score ranges from 12 to 60, with higher scores indicating a higher degree of walking impairment.
Modified Fatigue Impact Scale (MFIS) | Baseline
  To assess the perceived impact of fatigue in people with multiple sclerosis. The score ranges from 0 to 84, with higher scores indicating a higher degree of fatigue.
Beck Depression Inventory (BDI-II) | Baseline
  To monitor anxiety and depression. The score ranges from 0 to 63, with higher scores indicating a higher degree of depression.

OTHER OUTCOMES:
Expanded Disability Status Scale (EDSS) | Baseline
  The EDSS is a widely used scale for measuring the level of disability in individuals with multiple sclerosis (MS). Developed by Kurtzke in 1955, it assesses both the severity of neurological impairment and the degree of disability in various functional systems. The score ranges from 0 to 10, with higher scores indicating a higher degree of disability.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Università di Genova, Genova
  - IRCCS Santa Maria Nascente - Fondazione Don Carlo Gnocchi, Milan
  - Università degli Studi di Milano, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prosperini L, Di Filippo M. Beyond clinical changes: Rehabilitation-induced neuroplasticity in MS. Mult Scler. 2019 Sep;25(10):1348-1362. doi: 10.1177/1352458519846096. PMID 31469359
- [Background] Cattaneo D, Ferrarin M, Frasson W, Casiraghi A. Head control: volitional aspects of rehabilitation training in patients with multiple sclerosis compared with healthy subjects. Arch Phys Med Rehabil. 2005 Jul;86(7):1381-8. doi: 10.1016/j.apmr.2004.12.029. PMID 16003668
- [Background] Bonilauri A, Sangiuliano Intra F, Pugnetti L, Baselli G, Baglio F. A Systematic Review of Cerebral Functional Near-Infrared Spectroscopy in Chronic Neurological Diseases-Actual Applications and Future Perspectives. Diagnostics (Basel). 2020 Aug 12;10(8):581. doi: 10.3390/diagnostics10080581. PMID 32806516